CLINICAL TRIAL: NCT02076672
Title: Investigation of the Anti-Cancer Activity of Artichoke Extract in an Asbestos-Exposed Population (The ABOCA Phase II Trial)
Brief Title: Investigation of the Anti-Cancer Activity of Artichoke Extract in an Asbestos-Exposed Population
Acronym: ABOCA1
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ontario Clinical Oncology Group (OCOG) (Other)
Collaborators: Aboca Spa Societa' Agricola (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: OCOG-2013-ABOCA1
Record Dates: First submitted 2014-02-24; First posted 2014-03-03 (Estimated); Last update posted 2021-07-13 (Actual); Status verified 2021-07

CONDITIONS: Asbestos Exposure
Keywords: prevention; non-malignant asbestos-related disease; benign pleural disease; asbestosis
MeSH Terms: conditions — Asbestosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Artichoke WPC (Experimental): Artichoke WPC 500 mg capsules. Dose = 1000 mg (2 - 500 mg capsules) just before breakfast and 1000 mg (2 - 500 mg capsules) before dinner. Duration: daily for a period of 90 days.
  Interventions: Drug: Artichoke WPC

INTERVENTIONS:
Drug: Artichoke WPC — Artichoke WPC 500 mg capsules. Dose = 1000 mg (2 - 500 mg capsules) just before breakfast and 1000 mg (2 - 500 mg capsules) before dinner. Duration: daily for a period of 90 days.

SUMMARY:
This is a single-arm phase II trial to assess the biological activity (in a sub-cohort using a Simon two-stage Phase II design) and toxicity of Artichoke Whole Phytocomplex Concentrate (WPC). The objective of the study is to explore the potential for a non-toxic phytocomplex extract from the artichoke plant as a chemoprevention agent.

DETAILED DESCRIPTION:
In individuals exposed to asbestos and affected with asbestosis or asbestos-related benign pleural disease, and therefore at increased risk of mesothelioma, the investigators will evaluate whether the treatment with the commercially-available Artichoke Whole Phytocomplex Concentrate (Artichoke WPC) for 90 days will decrease mesothelin serum levels.

Although the investigators have general information on toxicity in humans, the investigators will monitor and assess the potential toxicity of Artichoke WPC in this patient population.

In addition to mesothelin, the investigators plan to evaluate the effects of Artichoke WPC on serum microRNAs (miRNAs). The use of miRNAs as minimally-invasive biomarkers has opened new opportunities for the diagnosis of cancer. A number of studies have addressed the potential association of disregulated miRNA profiling and benign asbestos-related disease and mesothelioma. Thus, the investigators will evaluate serum miRNA profiling before and after treatment with Artichoke WPC.

ELIGIBILITY:
Inclusion Criteria:

1. Asbestosis (defined as diffuse lung scarring based on increased profusion of interstitial fibrosis)
2. Benign pleural disease (defined as thickening or fibrotic plaques on pleural surfaces of the lung bilaterally)

Exclusion Criteria:

1. Prior systemic chemotherapy, radiation therapy or both.
2. A current or previous history of primary malignancy.
3. Known allergy to artichoke.
4. Known bile duct obstruction.
5. Known pregnancy or lactating women.
6. Known psychiatric illness/social situations that would limit study compliance.
7. Receiving any other investigational agents.
8. Inability to understand or unable to provide written informed consent.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2019-11-05 (Actual); Primary Completion 2020-04-28 (Actual); Study Completion 2020-04-28 (Actual)

PRIMARY OUTCOMES:
Efficacy outcome | 90 days post last subject recruitment
  The primary efficacy outcome is based on the reduction in serum concentration levels of mesothelin, measured at baseline and at the end of the intervention for subjects in the efficacy sub-cohort (i.e. for subjects who had elevated mesothelin levels at baseline). A positive outcome will be declared if the biomarker shows a reduction of 25% or more of its baseline value over the 90-day treatment period. For each study subject, mesothelin serum levels for both the baseline and final blood draws will be determined at the same time and in the same batch. This will assist in minimizing the technical variability of the assessments.

SECONDARY OUTCOMES:
Safety outcome | Day 45 and Day 90
  At the Day 45 and Day 90 visits, adverse reactions will be reported and graded according to the NCI CTCAE Version 4.03.

CONTACTS AND LOCATIONS:
Overall Officials: Paola Muti, Principal Investigator — McMaster University
Locations (1):
- St. Joseph's Hospital, Firestone Institute, Hamilton, Ontario, Canada

REFERENCES:
- [Derived] Muti P, Sacconi A, Pulito C, Orlandi G, Donzelli S, Morrone A, Jiulian J, Cox GP, Kolb M, Pond G, Kavsak P, Levine MN, Blandino G, Strano S. Artichoke phytocomplex modulates serum microRNAs in patients exposed to asbestos: a first step of a phase II clinical trial. J Exp Clin Cancer Res. 2022 Aug 20;41(1):255. doi: 10.1186/s13046-022-02455-6. PMID 35987988